CLINICAL TRIAL: NCT06862739
Title: Glycemic Control with Triple Pathway Approach Through Empagliflozin-Linagliptin-Metformin
Brief Title: Glycemic Control with Triple Pathway Approach Through Empagliflozin, Linagliptin and Metformin Combination
Acronym: GLYCO-3P
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nabiqasim Industries (Pvt) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NQ/DY/GLX/CT-001
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus; Type 2 DM
Keywords: Combination; empagliflozin; metformin; linagliptin; compliance; Hypoglycemic events; weight management; quality of life; treatment satisfaction; glycemic control; Type 2 DM
MeSH Terms: conditions — Diabetes Mellitus; Patient Compliance

STUDY DESIGN:
Intervention Model Description: 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glem-Lin MXR Single pill combination study (Other): Empagliflozin (25 mg) Linagliptin (5 mg) Metformin XR (1000 mg)
  once daily combination therapy
  Interventions: Combination Product: Empagliflozin+Linagliptin+Metformin

INTERVENTIONS:
Combination Product: Empagliflozin+Linagliptin+Metformin — Scarcity of local population data on triple drug combination's impact on compliance, efficacy and safety in diabetic patients

SUMMARY:
The efficacy and safety of a triple-pill combination therapy for advanced type 2 diabetes care. The study aims to assess the impact of 3 Oral Anti Diabetic (OAD) drugs on metabolic control, patient compliance, weight management, quality of life, diabetic treatment satisfaction and frequency of hypoglycemic events by combining them into a fixed-dose single pill.

DETAILED DESCRIPTION:
This study aims to demonstrate that a poly-pill approach combining metformin, linagliptin, and empagliflozin will provide an effective and safe treatment option for managing type 2 diabetes mellitus (T2DM). By focusing on the reduction of HbA1c levels and enhancing patients' quality of life, this simplified approach is expected to streamline medication regimens, reduce pill burden, and improve treatment adherence. Furthermore, the study anticipates that this combination therapy will positively influence weight management and lower the incidence of hypoglycemic events, addressing common challenges in T2DM management. As T2DM prevalence continues to rise, especially in low- and middle-income countries, the poly-pill strategy may offer significant benefits, promoting better compliance, affordable low-in-cost treatment, and facilitating improved long-term health outcomes. Through this research, the study intends to provide strong evidence supporting the poly-pill regimen as a viable and impactful option for global T2DM management.

ELIGIBILITY:
Inclusion criteria

1. Patients of any gender
2. Patients aged between 18-80 years
3. Patients having HbA1c 8 % or above
4. Patients diagnosed with type II diabetes (more than at least 06 months)
5. Patients already on at least 02 or more anti-diabetic agents
6. Patients not allergic to empagliflozin, linagliptin, or metformin

Exclusion criteria

1. Patients with age less than 18
2. Patients with Type-I diabetes
3. Patients having diabetes for less than 06 months
4. Patients on GLP-1 and GIP
5. Patients who are pregnant or lactating females
6. Patients with decompensated chronic liver disease (DCLD)
7. Patients with eGFR less than 30 ml
8. Patients with end-stage heart failure (NYHA Class 4)
9. Patients who are allergic to empagliflozin, linagliptin, or metformin
10. Patients who are not willing to consent
11. Patients who are unable to give medical history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c levels | 03 months, 06 months
  Metabolic control

SECONDARY OUTCOMES:
Change in scores of Quality of Life-Short Form "SF-36" questionnaire | 06 months
  Improvement in quality of life (before and after treatment)
Changes in Diabetic Treatment Satisfaction Questionnaire "DTSQ" | 06 months
  Diabetic treatment satisfaction level (before and after treatment)
Hypoglycemic events | 06 months
  Hypoglycemic events frequency and severity of hypoglycemic events
Changes in body weight | 03 and 06 months
  Increase or decrease in body weight

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Screening for Diabetes in Adults — https://pubmed.ncbi.nlm.nih.gov/29650090/
- See also: IDF diabetes atlas 2021 Pakistan's ranking — https://diabetesatlas.org/atlas/tenth-edition/
- See also: Health system performance for people with diabetes in LMICs — https://journals.plos.org/plosmedicine/article?id=10.1371/journal.pmed.1002751